CLINICAL TRIAL: NCT02592265
Title: Measuring Consequences of Disability for Patients With Multiple Sclerosis and Caregivers on Economic Burden and Social Participation.
Brief Title: Measuring Consequences of Disability for Patients With Multiple Sclerosis and Caregivers on Economic Burden
Acronym: ECOPASEP
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Université de Lille (Other); Région Nord-Pas de Calais, France (Other); La Ligue Française Contre la Sclérose en Plaques (Other); Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: RC-P0018
Record Dates: First submitted 2015-10-11; First posted 2015-10-30 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis; Physical Disability; Economic Burden; Social Interaction; Capability; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Financial Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to measure economic burden of Multiple Sclerosis (MS) from a new point of view that includes consequences of disability on Quality Of Life (QOL), social participation and capabilities of patients and caregivers. To the investigators' knowledge, there is currently no data including intangible costs related to caregivers and calculating the overall economic cost of Multiple Sclerosis, particularly, in France.

DETAILED DESCRIPTION:
The goal of this study is to evaluate prospectively the economic burden of Multiple Sclerosis (MS) in France by calculating direct costs (medical and non-medical) and indirect costs and by estimating consequences of MS on utility (QALY) of patients and caregivers in a societal perspective.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 or more
* Confirmed MS diagnosis (McDonald 2005)
* Defined type of MS according classification of Lublin and Reingold

Exclusion Criteria:

* Subject living in an institution
* Severe cognitive dysfunction preventing to answer questionnaire
* Subject already included in other clinical study (phase 1 to 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 230 patients in secondary and tertiary centers (8) affiliated to the regional supportive care network (GSEP) in north of France.
Sampling Method: Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2012-10; Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Annual average total health care cost of the Multiple Sclerosis by patient | 1 year
  Global cost of Multiple Sclerosis considering direct medical and non-medical costs as well as the indirect and intangible costs associated to the patient-caregiver

SECONDARY OUTCOMES:
Score of social participation | 1 year
  Correlation between the score of social participation and health care costs of the disease will be determined
Validity of life quality measurement EQ-5D | 1 year
  The EQ-5D index is a generic measure of health status that provides a simple descriptive profile and a single index value that can be used in the clinical and economic evaluation of health care
Utilities measured by the Short Form-6D (SF-6D) | 1 year
  The SF-6D is a utility index based on a descriptive system composed of 11 items from six dimensions of the SF-36: physical functioning, role limitations, social functioning, pain, mental functioning and vitality.
QALY | 1 year
  Health related quality in life will be measured as Quality adjusted life years (QALY)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud KWIATKOWSKI, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille; Amélie LANSIAUX, Study Director — Groupement des Hôpitaux de l'Institut Catholique de LilleGroupement des Hôpitaux de l'Institut Catholique de Lille